CLINICAL TRIAL: NCT05690555
Title: A Randomized Trial Comparing Perioperative Pelvic Floor Physical Therapy to Current Standard of Care in Transgender Women Undergoing Vaginoplasty for Gender Affirmation
Brief Title: Pelvic Floor Physical Therapy vs Standard Care in Transgender Women Undergoing Vaginoplasty for Gender Affirmation
Acronym: FLOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-917
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT) (Experimental): If patients were randomized into the PFPT arm, they were further randomized into the following sub-arms: Preoperative and Postoperative PFPT
  Interventions: Other: Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT)
- Postoperative Pelvic Floor Physical Therapy (PFPT) (Active Comparator): Patients will present to see the physical therapist 3 weeks postoperatively. The following interventions will be performed: Subjective assessment of bowel and bladder function. Visual and external palpation and assessment of external pelvic floor region. Intravaginal pelvic floor assessment. Pelvic floor muscle dynamics and coordination assessment. Review of pelvic floor anatomy and function.
  Interventions: Other: Postoperative PFPT
- No Pelvic Floor Physical Therapy (PFPT) (Active Comparator): Patients were not assigned to physical therapy.
  Interventions: Other: No Pelvic Floor Physical Therapy (PFPT)

INTERVENTIONS:
Other: Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT) — Patients will present to see the physical therapist 3 weeks and 6 weeks postoperatively. The following interventions will be performed:
  3 weeks:
  * Subjective assessment of bowel and bladder function
  * Visual and external palpation and assessment of external pelvic floor region
  * Intravaginal pelvic floor assessment
  * Pelvic floor muscle dynamics and coordination assessment
  * Instruction of pelvic floor coordination and lengthening
  * Discussion of dilator program and progression
  * Home program with instructions
    6 weeks:
  * External scar assessment and treatment if tissue healing allows
  * Instruction to patient of scar mobilizations
  * Intravaginal pelvic floor assessment and treatment if indicated
  * Review of pelvic floor lengthening and coordination
  * Review and progression of dilator program if appropriate
  * Assessment of current bowel/bladder symptoms; home program and instructions to address these symptoms
  Arms: Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT)
Other: No Pelvic Floor Physical Therapy (PFPT) — Patients will present to see the physical therapist 3 weeks postoperatively. The following interventions will be performed:
  Subjective assessment of bowel and bladder function. Visual and external palpation and assessment of external pelvic floor region. Intravaginal pelvic floor assessment. Pelvic floor muscle dynamics and coordination assessment. Review of pelvic floor anatomy and function.
  Arms: No Pelvic Floor Physical Therapy (PFPT)
Other: Postoperative PFPT — Preoperative Diaphragmatic breathing Discuss dilator positioning/introduce dilator program External pelvic floor assessment Teach pelvic floor coordination Current bowel/bladder symptoms; home program and instructions 3 weeks Assessment of bowel and bladder function Visual and external palpation and assessment of external pelvic floor region Intravaginal pelvic floor assessment Pelvic floor muscle dynamics and coordination assessment Instruction of pelvic floor coordination and lengthening Discussion of dilator program and progression Home program with instructions 6 weeks External scar assessment and treatment if tissue healing allows Instruction to patient of scar mobilizations Intravaginal pelvic floor assessment and treatment if indicated Review of pelvic floor lengthening and coordination Review and progression of dilator program if appropriate Current symptoms; home program and instructions
  Arms: Postoperative Pelvic Floor Physical Therapy (PFPT)

SUMMARY:
Currently, perioperative pelvic floor physical therapy (PFPT) is not standard of care for all patients who undergo vaginoplasty surgery. While some practices have implemented these new programs, and the above data exist on outcomes associated with perioperative PFPT in transgender women undergoing vaginoplasty, no study has compared implementation of perioperative PFPT to routine care (no perioperative PFPT). Therefore, the primary objective of this study was to compare the effectiveness of postoperative PFPT compared to no PFPT in transgender women undergoing vaginoplasty surgery for gender affirmation. Secondary objectives of the study are 1) to describe the incidence of preoperative pelvic floor dysfunction in transgender women undergoing PFPT and 2) to compare the effectiveness of postoperative PFPT alone to pre- and postoperative PFPT in these patients.

DETAILED DESCRIPTION:
This was a randomized double-blind study. Both subjects and the surgeon performing the surgery as well as the personnel administering questionnaires to patients postoperatively were blinded to the randomization.

Recruitment, Enrollment and Randomization

Patients scheduled to undergo vaginoplasty surgery at Cleveland Clinic Main campus were approached about voluntary participation in this study. This occurred over the phone approximately one to three months before their scheduled surgery. Patients who agreed to participate were sent a consent form via the mail and were asked to sign consent in person. Enrollment and randomization occurred following informed consent. All patients were given a copy of their signed and dated consent.

Once enrolled, patients were randomized into one of two groups:

* Postoperative PFPT
* No Postoperative PFPT

If patients were randomized into the Postoperative PFPT arm, they were further randomized into the following sub-arms:

* Postoperative PFPT alone
* Preoperative and Postoperative PFPT

Surgery:

All patients underwent vaginoplasty surgery by a single surgeon in a standard fashion. The neovaginal cavity was created using the same technique across all patients. Postoperative care was routine and the same for all patients.

Postoperative Pelvic Floor Physical Therapy:

There was three possible PFPT regimens. All PT regimens were performed by the same two physical therapists, trained in the management of patients who have undergone vaginoplasty surgery.

1. No PFPT Patients were present to see the physical therapist 3 weeks postoperatively. The following interventions were performed: Subjective assessment of bowel and bladder function. Visual and external palpation and assessment of external pelvic floor region. Intravaginal pelvic floor assessment. Pelvic floor muscle dynamics and coordination assessment. Review of pelvic floor anatomy and function.
2. Postoperative PFPT Only

Patients presented to the physical therapist 3 weeks and 6 weeks postoperatively. The following interventions were performed:

3 weeks:

* Subjective assessment of bowel and bladder function
* Visual and external palpation and assessment of external pelvic floor region
* Intravaginal pelvic floor assessment
* Pelvic floor muscle dynamics and coordination assessment
* Instruction of pelvic floor coordination and lengthening
* Discussion of dilator program and progression
* Home program with instructions

  6 weeks:
* External scar assessment and treatment if tissue healing allows
* Instruction to patient of scar mobilizations
* Intravaginal pelvic floor assessment and treatment if indicated
* Review of pelvic floor lengthening and coordination
* Review and progression of dilator program if appropriate
* Assessment of current bowel/bladder symptoms; home program and instructions to address these symptoms

  3) Preoperative PFPT and Postoperative PFPT:

Patients presented to see the physical therapist 3 weeks before surgery, 3 weeks and 6 weeks postoperatively. The following interventions were performed:

Preoperative:

* Diaphragmatic breathing
* Discuss dilator positioning/introduce dilator program
* External pelvic floor assessment
* Teach pelvic floor coordination
* Assessment of current bowel/bladder symptoms; home program and instructions to address these symptoms

  3 weeks:
* Subjective assessment of bowel and bladder function
* Visual and external palpation and assessment of external pelvic floor region
* Intravaginal pelvic floor assessment
* Pelvic floor muscle dynamics and coordination assessment
* Instruction of pelvic floor coordination and lengthening
* Discussion of dilator program and progression
* Home program with instructions

  6 weeks:
* External scar assessment and treatment if tissue healing allows
* Instruction to patient of scar mobilizations
* Intravaginal pelvic floor assessment and treatment if indicated
* Review of pelvic floor lengthening and coordination
* Review and progression of dilator program if appropriate
* Assessment of current bowel/bladder symptoms; home program and instructions to address these symptoms

Study Questionnaires & Exams:

All patients were administered questionnaires preoperatively and 12 weeks postoperatively. The following questionnaires were administered:

Preoperatively:

* CRAD-8 and UDI-6
* PFIQ-7

Postoperatively 1 week (at the time of routine dilation teaching):

• Vaginal length (routine exam)

Postoperatively 12 weeks:

* CRAD-8 and UDI-6
* PFIQ-7
* PGI-I
* Ease of Passing Dilator (VAS 0-10)
* Pain with Dilation (VAS 0-10)
* Largest dilator size used
* Vaginal length (routine exam)

Cross-Over Treatment:

Any patients in the No PFPT arm who were determined to have pelvic floor dysfunction or symptoms that may have benefitted from PFPT referral, were referred after the 12-week mark. Any patient in one of the PFPT arms who was determined to still need PFPT for persistent pelvic floor dysfunction or symptoms were referred for continued care.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age
* Patients scheduled for full-depth vaginoplasty surgery

Exclusion Criteria:

* Inability to speak or comprehend the English language
* Patients scheduled for no-depth vaginoplasty surgery
* Patients who have undergone previous PFPT
* Patients who are s/p prostatectomy or treatment for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women are individuals who were assigned male at birth (are biologically male), but identify as female.
Enrollment: 37 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Ferrando, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Postoperative Pelvic Floor Physical Therapy (PFPT): Pelvic Floor Physical Therapy (PFPT): Patients will present to see the physical therapist 3 weeks and 6 weeks postoperatively. The following interventions will be performed:
  3 weeks:
  * Subjective assessment of bowel and bladder function
  * Visual and external palpation and assessment of external pelvic floor region
  * Intravaginal pelvic floor assessment
  * Pelvic floor muscle dynamics and coordination assessment
  * Instruction of pelvic floor coordination and lengthening
  * Discussion of dilator program and progression
  * Home program with instructions
    6 weeks:
  * External scar assessment and treatment if tissue healing allows
  * Instruction to patient of scar mobilizations
  * Intravaginal pelvic floor assessment and treatment if indicated
  * Review of pelvic floor lengthening and coordination
  * Review and progression of dilator program if appropriate
  * Assessment of current bowel/bladder symptoms; home program and instructions to address these symptoms
- No Postoperative Pelvic Floor Physical Therapy (PFPT): Patients will present to see the physical therapist 3 weeks postoperatively. The following interventions will be performed: Subjective assessment of bowel and bladder function. Visual and external palpation and assessment of external pelvic floor region. Intravaginal pelvic floor assessment. Pelvic floor muscle dynamics and coordination assessment. Review of pelvic floor anatomy and function.
  No Pelvic Floor Physical Therapy (PFPT): Patients will present to see the physical therapist 3 weeks postoperatively. The following interventions will be performed:
  Subjective assessment of bowel and bladder function. Visual and external palpation and assessment of external pelvic floor region. Intravaginal pelvic floor assessment. Pelvic floor muscle dynamics and coordination assessment. Review of pelvic floor anatomy and function.
  Cross-over Treatment: Any patients in the No PFPT arm who are determined to have pelvic floor dysfunction or symptoms that may benefit from PFPT referral, will be referred after the 12-week mark. Any patient in one of the PFPT arms who is determined to still need PFPT for persistent pelvic floor dysfunction or symptoms will be referred for continued care.
- Pre and Postoperative Pelvic Floor Physical Therapy (PFPT): Pelvic Floor Physical Therapy (PFPT): Patients will present to see the physical therapist within 4 weeks preceding surgery and 3 weeks and 6 weeks postoperatively. The following interventions will be performed:
  Preoperative:
  Teaching about the pelvic floor and breathing exercises
  3 weeks:
  * Subjective assessment of bowel and bladder function
  * Visual and external palpation and assessment of external pelvic floor region
  * Intravaginal pelvic floor assessment
  * Pelvic floor muscle dynamics and coordination assessment
  * Instruction of pelvic floor coordination and lengthening
  * Discussion of dilator program and progression
  * Home program with instructions
    6 weeks:
  * External scar assessment and treatment if tissue healing allows
  * Instruction to patient of scar mobilizations
  * Intravaginal pelvic floor assessment and treatment if indicated
  * Review of pelvic floor lengthening and coordination
  * Review and progression of dilator program if appropriate
  * Assessment of current bowel/bladder symptoms; home program and instructions to address these symptoms
Period: Overall Study
Arm/Group | Postoperative Pelvic Floor Physical Therapy (PFPT) | No Postoperative Pelvic Floor Physical Therapy (PFPT) | Pre and Postoperative Pelvic Floor Physical Therapy (PFPT)
Started | 10 | 17 | 10
Completed | 10 | 17 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Postoperative Pelvic Floor Physical Therapy (PFPT) | No Postoperative Pelvic Floor Physical Therapy (PFPT) | Pre and Postoperative Pelvic Floor Physical Therapy (PFPT) | Total
Number analyzed (Participants) | 10 | 17 | 10 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 17 | 10 | 37
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33 (7) | 28 (14) | 36 (15) | 32.3 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 17 | 10 | 37
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 5
  White | 9 | 14 | 9 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 17 | 10 | 37

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Ease of Dilation
Description: VAS 0-10 is a validated 10 item questionnaire. Responses to each question are scored on a 10-point Likert scale, ranging from 0 (no pain) to 10 (worst pain). A response of 10 is considered to be a worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT): Patients who were further randomized to also undergo a preoperative PFPT visit were taught about diaphragmatic breathing at this visit, they were introduced to the postoperative dilator program, underwent an external pelvic floor assessment, and were taught pelvic floor coordination.
Arm/Group | Postoperative Pelvic Floor Physical Therapy (PFPT) | No Postoperative Pelvic Floor Physical Therapy (PFPT) | Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT)
Number analyzed (Participants) | 10 | 17 | 10
units on a scale | 6.6 (1.9) | 7.4 (1.7) | 8.0 (0.8)

2. Post Hoc Outcome: Severity of Pelvic Floor Dysfunction Based on PGI-I
Description: The Patient Global Impression of Improvement (PGI-I) is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1 (very much better) to 7 (very much worse). A score of 7 is considered to be a worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Postoperative Pelvic Floor Physical Therapy (PFPT) | No Postoperative Pelvic Floor Physical Therapy (PFPT) | Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT)
Number analyzed (Participants) | 10 | 17 | 10
units on a scale | 1.4 (0.7) | 1.65 (1.49) | 1.9 (1.3)

3. Post Hoc Outcome: Mean Difference in CRADI-8 Score
Description: Colorectal-Anal Distress Inventory (CRADI-8) provides a symptom inventory (no or yes) and if yes (to measure the degree of bother and distress) caused by the broad array of pelvic floor symptoms, in particular colorectal-anal distress. Responses to the eight questions are scored on a 4-point Likert scale, ranging 1 (not at all) to 4 (quite a bit). The scale scores are found individually by calculating the mean value of their corresponding questions and then multiplying by 25 to obtain a value that ranges from 0 to 100. The reported outcome for this trial is the mean difference in score. A higher CRADI-8 score indicates a greater level of disability. It reflects more significant challenges in daily activities and functioning. A score of 100 is considered to be a worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Postoperative Pelvic Floor Physical Therapy (PFPT) | No Postoperative Pelvic Floor Physical Therapy (PFPT) | Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT)
Number analyzed (Participants) | 10 | 17 | 10
units on a scale | -0.6 (3.69) | -3.00 (7.37) | -1.9 (7.58)

4. Post Hoc Outcome: Mean Difference UDI-6 Score
Description: Urinary Distress Inventory (UDI-6) - The UDI-6 is a 6-item questionnaire. Each item is scored on a scale of 0 to 3, with 0 being "not at all" and 3 being "greatly". The average score is calculated and multiplied by 33 1/3 to give a score on a scale of 0 to 100. A higher score indicates a higher level of disability. The outcome measure reported in this trial is the mean difference in scores pre- and post-intervention. A higher UDI-6 score indicates a greater level of disability. It reflects more significant challenges in daily activities and functioning. A score of 100 is considered to be a worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Postoperative Pelvic Floor Physical Therapy (PFPT) | No Postoperative Pelvic Floor Physical Therapy (PFPT) | Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT)
Number analyzed (Participants) | 10 | 17 | 10
units on a scale | -1.5 (14.6) | -1.41 (7.14) | -6.5 (32.02)

5. Post Hoc Outcome: Mean Difference PFIQ-7-Bladder Score
Description: The Pelvic Floor Impact Questionnaire-7 (PFIQ-7) is a seven-question survey that measures the impact of pelvic floor disorders on quality of life, daily activities, and emotional health. The PFIQ-7 is scored on a scale of 0-300. The mean of each of the three scales is calculated, ranging from 0-3. Each mean is multiplied by 100 and then divided by 3. The scale scores are added together to get the total PFIQ-7 score. The reported outcome measure in this trial is the mean difference in this score pre- and post-intervention. A higher PFIQ-7 score indicates a greater level of disability. It reflects more significant challenges in daily activities and functioning. A score of 300 is considered to be a worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Postoperative Pelvic Floor Physical Therapy (PFPT) | No Postoperative Pelvic Floor Physical Therapy (PFPT) | Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT)
Number analyzed (Participants) | 10 | 17 | 10
units on a scale | 6.7 (22.99) | -1.64 (10.45) | -4.8 (18.4)

6. Post Hoc Outcome: Mean Difference in PFIQ-7-Rectum Score
Description: The Pelvic Floor Impact Questionnaire-7 (PFIQ-7) is a seven-question survey that measures the impact of pelvic floor disorders on quality of life, daily activities, and emotional health. The PFIQ-7 is scored on a scale of 0-300. The mean of each of the three scales is calculated, ranging from 0-3. Each mean is multiplied by 100 and then divided by 3. The scale scores are added together to get the total PFIQ-7 score. The reported outcome measure in this trial is the mean difference in this score pre- and post-intervention. A score of 300 is considered to be a worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Postoperative Pelvic Floor Physical Therapy (PFPT) | No Postoperative Pelvic Floor Physical Therapy (PFPT) | Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT)
Number analyzed (Participants) | 10 | 17 | 10
units on a scale | 6.2 (23.21) | -3.17 (11.31) | 0.5 (3.69)

7. Post Hoc Outcome: Mean Difference in PFIQ-7-Vagina Score
Description: as for outcome 5
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Postoperative Pelvic Floor Physical Therapy (PFPT) | No Postoperative Pelvic Floor Physical Therapy (PFPT) | Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT)
Number analyzed (Participants) | 10 | 17 | 10
units on a scale | 6.3 (27.65) | 5.65 (18.18) | 3.5 (15.0)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- No Postoperative Pelvic Floor Physical Therapy (PFPT): No Pelvic Floor Physical Therapy (PFPT): Patients will present to see the physical therapist 3 weeks postoperatively. The following interventions will be performed:
  Subjective assessment of bowel and bladder function. Visual and external palpation and assessment of external pelvic floor region. Intravaginal pelvic floor assessment. Pelvic floor muscle dynamics and coordination assessment. Review of pelvic floor anatomy and function.
Arm/Group | Postoperative Pelvic Floor Physical Therapy (PFPT) | No Postoperative Pelvic Floor Physical Therapy (PFPT) | Preoperative and Postoperative Pelvic Floor Physical Therapy (PFPT)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/17 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/17 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/17 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT05690555/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT05690555/ICF_001.pdf